CLINICAL TRIAL: NCT06750809
Title: A Prospective Post-Market Multicenter Randomized Controlled Clinical Study to Investigate Clinical Outcomes and Associated Costs When PermeaDerm is Used as Temporary Dressing for the Management of Surgical Wounds
Brief Title: Randomized Controlled Trial to Investigate Clinical Outcomes and Associated Costs When PermeaDerm is Used as Temporary Dressing for Surgical Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP012
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Surgical Wound; Trauma Wound; Autografts; Partial-thickness Burn; Partial Thickness Wounds
Keywords: Skin graft, surgical wound, trauma wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PermeaDerm Temporary Biosynthetic Wound Matrix (Experimental)
  Interventions: Device: PermeaDerm Biosynthetic Wound Matrix
- Frozen Human Cadaveric Allograft (FHCA) (Experimental)
  Interventions: Device: Frozen Human Cadaveric Allograft (FHCA)

INTERVENTIONS:
Device: PermeaDerm Biosynthetic Wound Matrix — Study participants randomized (1:1) to this arm will receive PermeaDerm Biosynthetic Wound Matrix prior to skin graft.
  Arms: PermeaDerm Temporary Biosynthetic Wound Matrix
Device: Frozen Human Cadaveric Allograft (FHCA) — Study participant randomized (1:1) to this arm will receive Frozen Human Cadaveric Allograft (FHCA) prior to skin graft.
  Arms: Frozen Human Cadaveric Allograft (FHCA)

SUMMARY:
The goal of this study is to compare the cost and clinical outcomes for two temporary dressings (Allograft and PermeaDerm) used in patients that need a skin graft to heal their wound. The researchers will review cost and other treatment results including how well both temporary dressings attach to the skin, how prepared the wound bed is to receive a skin graft, how long it takes for the skin to be ready to receive a skin graft, how well the skin graft takes and any complications. Patients will first have the temporary dressing applied to their wound, then a few days later, a skin graft will be performed. Patients will have photos of their wounds taken throughout the study including at all the clinic check-ups with the last check-up occurring about 8 weeks after treatment.

DETAILED DESCRIPTION:
This is a prospective two-arm randomized multicenter controlled study to evaluate the clinical outcomes and economic impact of PermeaDerm and frozen human cadaveric allograft (FHCA) when they are used as a temporary dressing on surgical wounds where autografting is clinically indicated.

Patients hospitalized within 3 days of injury with a surgical wound up to 30% (inclusive) total body surface area (TBSA) will be considered for participation in this study.

Patients will undergo surgical excision within five days post-injury and will be randomly assigned (1:1) to receive PermeaDerm or FHCA as a temporary dressing. One contiguous area will be selected by the investigator as the study treatment area. Any other areas that require a temporary dressing must be dressed per the randomization.

In addition to economic impact, the two temporary dressings will be compared with respect to adherence, wound bed preparation, time to autografting, graft take, and safety-related adverse events.

Following placement of the temporary dressing, investigators will evaluate the wound every 2-3 days. The temporary dressing may be replaced, per the randomization, as clinically indicated. When the study area is ready for autografting, the temporary dressing will be removed, and the study area will be autografted per the investigative site's standard of care. The donor area(s) may be dressed in PermeaDerm or the investigative site's standard of care.

Post-autografting, subjects will be followed for 8 weeks. Treatment-related and serious adverse events will be reported through the duration of the study. At all visits, subjects' study treatment areas and donor sites that are dressed in PermeaDerm will be documented using digital photography.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible for participation:

1. The patient's wound requires temporary dressing coverage after surgical excision and prior to autografting.
2. The patient has a surgical wound up to 30% (inclusive) total body surface area (TBSA).
3. The study area is a contiguous area. If the patient has other areas (non-study treatment area) that require temporary dressing, these areas must also be dressed according to the randomization.
4. The patient is hospitalized within 3 days of injury.
5. The surgical excision occurs within 5 days post-injury.
6. The patient (or parent/guardian/legally authorized representative) is willing and able to comply with all study procedures and visit schedule.
7. The patient (or parent/guardian/legally authorized representative) agrees to abstain from any other treatment of the study area or enrollment in another interventional clinical trial for the duration of his/her participation in the study (8 weeks post-autografting).
8. In the opinion of the investigator, the patient (or parent/guardian/legally authorized representative) must be able to:

   1. Understand the full nature and purpose of the study, including possible risks and adverse events,
   2. Understand instructions, and
   3. Provide voluntary written informed consent.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible for participation:

1. The study area has received prior surgical intervention.
2. The patient is currently using medications or treatments such as systemic corticosteroids, chemotherapy, or immunosuppressants, that in the investigator's opinion may compromise patient safety or trial objectives.
3. Clinical signs of wound infection at study area that in the investigator's opinion may compromise patient safety or trial objectives.
4. The patient has any of the following

   1. morbid obesity (BMI >40),
   2. immunodeficiency,
   3. venous insufficiency/PVD of the lower extremities (when study area is also in this location),
   4. chronic malnourishment,
   5. inhalation injury (>Grade 1 based on AIS grading scale),
   6. current abuser of alcohol and/or illicit drugs based upon medical history and/or lab results,
   7. diabetes mellitus with HbA1c >9.0%, and/or
   8. advanced renal disease (eGFR <59) or liver disease (LFTs >2.5 times the upper limit).
5. The patient has any another condition, that in the investigator's opinion may compromise patient safety or the trial objectives.
6. The patient is unable to understand English or Spanish.
7. The patient has a known hypersensitivity to bovine-derived collagen materials, porcine, aloe vera materials, or contraindications to the frozen human cadaveric allograft.
8. The patient's life expectancy is less than 1 year.

   -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of Cost per Total Body Surface Area (TBSA) | 8 weeks post treatment.
  The reduction of cost per TBSA when PermeaDerm is used as a temporary dressing. The reduction in cost is hypothesized to be superior for PermeaDerm as compared to FHCA.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Valleywise Health, Phoenix, Arizona
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Grady Memorial, Atlanta, Georgia
  - Univ of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Univ of Louisville Burn Center, Louisville, Kentucky
  - University Medical Center, New Orleans, Louisiana
  - University of Rochester, Rochester, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Ohio State University, Columbus, Ohio
  - Regional One Firefighter's Burn Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No